CLINICAL TRIAL: NCT05644314
Title: Efficacy of Drug-Eluting Vertebral Artery Stenting Treatment for Atherosclerotic Vertebral Arteries Stenosis in Real-World Clinical Observations: a Prospective, Multicenter, Open-access, Single-arm Clinical Study
Brief Title: Efficacy of Drug-Eluting Vertebral Artery Stenting Treatment for Atherosclerotic Vertebral Arteries Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, jizhong, Associate chief physician, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-410
Record Dates: First submitted 2022-11-16; First posted 2022-12-09 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Stroke; Vertebral Artery Stenosis
MeSH Terms: conditions — Ischemic Stroke; Vertebrobasilar Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with vertebral atherosclerotic stenosis requiring stent implantation (Experimental): Referring to "the 2015 Chinese Guidelines for Endovascular Interventional Treatment of Ischemic Cerebrovascular Disease", "the 2015 Symptomatic Atherosclerotic Sclerotic vertebral artery initiation stenosis: Chinese expert consensus" and "Subclavian/extracranial vertebral artery stenosis: Chinese expert consensus" in 2019 and other guidelines and expert consensus for the diagnosis of symptomatic vertebral artery atherosclerotic stenosis ≥ 50% and non-symptomatic vertebral artery atherosclerotic stenosis ≥ 70% in patients.
  Interventions: Device: The drug-eluting stent

INTERVENTIONS:
Device: The drug-eluting stent — Vertebral artery drug-eluting stents Maurora® was approved for marketing in 2020 and has been shown to be effective in reducing restenosis in clinical trials.

SUMMARY:
This is a prospective, multi-center, open-access, single-arm trial to observe the real-world clinical efficacy of drug-eluting vertebral artery stenting system treatment for Atherosclerotic Vertebral Arteries Stenosis. Patients will be followed at 30 days, 6, and 12 months post-procedure and annually for 1 year within 3 years.

DETAILED DESCRIPTION:
Stroke has been one of the most important causes of disability and death worldwide today. Ischemic stroke accounts for more than 50% of these strokes. The results of epidemiological surveys show that in 2018, more than 3 million new strokes occurred each year in China. In 2018, more than 3 million people suffered from a stroke, and more than 2 million people died from a stroke. Studies show that about 25% to 40% of transient ischemic attacks (TIA) or strokes occur in the posterior circulation. The subclavian and vertebral arteries are important blood vessels in the posterior circulation and are important original sites for ischemic strokes in the posterior circulation. About 20% of strokes in the posterior circulation are caused by extracranial vertebral artery stenosis (ECVAS). Endovascular intervention is the recommended treatment for ECVAS. It is effective in promoting the perfusion of brain tissue in the area of the responsible artery, thereby reducing the risk of stroke recurrence, improving neurological prognosis, and reducing symptoms. The drug-eluting stent is effective in reducing the incidence of postoperative restenosis (ISR), thus further reducing the long-term risk of stroke. Vertebral artery drug-eluting stents Maurora® was approved for marketing in 2020 and has been shown to be effective in reducing restenosis in clinical trials. The purpose of this study is to further investigate its long-term effectiveness in treating vertebral artery stenosis in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender is not limited;
2. Patients with medically prescribed rapamycin drug-eluting vertebral artery stent systems;
3. Patients and family members fully understand the trial's purpose, voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Unable to receive dual antiplatelet therapy due to known disease, or severe coagulation abnormalities, severe infections that are not controlled, severe systemic disease, uncontrollable hypertension, and contraindicated for surgery;
2. With an aneurysm that cannot be treated earlier or simultaneously or is not suitable for surgery;
3. Gastrointestinal disease with active bleeding;
4. Previous myocardial infarction or large-scale cerebral infarction within 2 weeks;
5. Known contraindications to heparin, rapamycin, anesthesia, and contrast agents;
6. Life expectancy less than 12 months;
7. the investigator judged patients to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinical ischemic events | within 1 year
  Examples of clinical cerebral ischemic events: TIA or ischemic stroke event in the blood supply area of the target lesion

SECONDARY OUTCOMES:
Clinical Success Rate | within 1 year after surgery
  Successful arrival and release of the stent in the target lesion with complete coverage of the lesion and residual stenosis <30%, no major adverse events (MAE).
Major adverse event (MAE) incidence | 1 month, 6 months, 12 months, 2 and 3 years
  Major adverse events (MAE) include all-cause death, any type of stroke (ischemic/hemorrhagic stroke) within 30 days of surgery, TIA or ischemic stroke in the target lesion supply area within 1 year, clinically driven target lesion revascularization (CD-TVL), thrombotic event.
Incidence of bleeding events | 30 days and 1 year
  Access or non access site bleeding
Incidence of in-stent restenosis | within 1 year
  Restenosis: in-stent stenosis rate ≥50% on imaging
Changes in the modified Rankin scale (mRS) scores | 1 month, 6 months, 12 months, 2 and 3 years
  ability to perform daily living，mRS scores ranges 0-6 ， the more score the more severe outcome
Change in NIHSS scores | 1 month, 6 months, 12 months, 2 and 3 years
  NIHSS scores for neurological deficits
Correlation of risk factors with the occurrence of major adverse events | 1 month, 6 months, 12 months, 2 and 3 years
  Major adverse events (MAE) include all-cause death, any type of stroke (ischemic/hemorrhagic stroke) within 30 days of surgery, TIA or ischemic stroke in the target lesion supply area within 1 year, clinically driven target lesion revascularization (CD-TVL), thrombotic event.
Correlation of risk factors with the occurrence of restenosis | 1 month, 6 months, 12 months, 2 and 3 years
  Thrombosis in study stents
Evaluation of clinical use for relative contraindications | 1 month, 6 months, 12 months, 2 and 3 years
  Evaluation of clinical cerebral ischemic events: TIA or ischemic stroke event in the blood supply area of the target lesion for contraindications patients

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Ji, PHD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The study is proceeding.

REFERENCES:
- [Result] Carrera E, Maeder-Ingvar M, Rossetti AO, Devuyst G, Bogousslavsky J; Lausanne Stroke Registry. Trends in risk factors, patterns and causes in hospitalized strokes over 25 years: The Lausanne Stroke Registry. Cerebrovasc Dis. 2007;24(1):97-103. doi: 10.1159/000103123. Epub 2007 May 23. PMID 17519551
- [Result] Marquardt L, Kuker W, Chandratheva A, Geraghty O, Rothwell PM. Incidence and prognosis of > or = 50% symptomatic vertebral or basilar artery stenosis: prospective population-based study. Brain. 2009 Apr;132(Pt 4):982-8. doi: 10.1093/brain/awp026. Epub 2009 Mar 17. PMID 19293244
- [Result] Caplan LR, Amarenco P, Rosengart A, Lafranchise EF, Teal PA, Belkin M, DeWitt LD, Pessin MS. Embolism from vertebral artery origin occlusive disease. Neurology. 1992 Aug;42(8):1505-12. doi: 10.1212/wnl.42.8.1505. PMID 1641144
- [Result] Gulli G, Marquardt L, Rothwell PM, Markus HS. Stroke risk after posterior circulation stroke/transient ischemic attack and its relationship to site of vertebrobasilar stenosis: pooled data analysis from prospective studies. Stroke. 2013 Mar;44(3):598-604. doi: 10.1161/STROKEAHA.112.669929. Epub 2013 Feb 5. PMID 23386676
- [Result] Gulli G, Khan S, Markus HS. Vertebrobasilar stenosis predicts high early recurrent stroke risk in posterior circulation stroke and TIA. Stroke. 2009 Aug;40(8):2732-7. doi: 10.1161/STROKEAHA.109.553859. Epub 2009 May 28. PMID 19478210
- [Result] Wang Y, Wang Y, Zhao X, Liu L, Wang D, Wang C, Wang C, Li H, Meng X, Cui L, Jia J, Dong Q, Xu A, Zeng J, Li Y, Wang Z, Xia H, Johnston SC; CHANCE Investigators. Clopidogrel with aspirin in acute minor stroke or transient ischemic attack. N Engl J Med. 2013 Jul 4;369(1):11-9. doi: 10.1056/NEJMoa1215340. Epub 2013 Jun 26. PMID 23803136
- [Result] Stayman AN, Nogueira RG, Gupta R. A systematic review of stenting and angioplasty of symptomatic extracranial vertebral artery stenosis. Stroke. 2011 Aug;42(8):2212-6. doi: 10.1161/STROKEAHA.110.611459. Epub 2011 Jun 23. PMID 21700936
- [Result] Markus HS, Harshfield EL, Compter A, Kuker W, Kappelle LJ, Clifton A, van der Worp HB, Rothwell P, Algra A; Vertebral Stenosis Trialists' Collaboration. Stenting for symptomatic vertebral artery stenosis: a preplanned pooled individual patient data analysis. Lancet Neurol. 2019 Jul;18(7):666-673. doi: 10.1016/S1474-4422(19)30149-8. Epub 2019 May 23. PMID 31130429
- [Result] Antoniou GA, Murray D, Georgiadis GS, Antoniou SA, Schiro A, Serracino-Inglott F, Smyth JV. Percutaneous transluminal angioplasty and stenting in patients with proximal vertebral artery stenosis. J Vasc Surg. 2012 Apr;55(4):1167-77. doi: 10.1016/j.jvs.2011.09.084. Epub 2011 Dec 28. PMID 22206680
- [Result] Langwieser N, Buyer D, Schuster T, Haller B, Laugwitz KL, Ibrahim T. Bare metal vs. drug-eluting stents for extracranial vertebral artery disease: a meta-analysis of nonrandomized comparative studies. J Endovasc Ther. 2014 Oct;21(5):683-92. doi: 10.1583/14-4713MR.1. PMID 25290797
- [Result] Lee JM, Park J, Kang J, Jeon KH, Jung JH, Lee SE, Han JK, Kim HL, Yang HM, Park KW, Kang HJ, Koo BK, Kim HS. Comparison among drug-eluting balloon, drug-eluting stent, and plain balloon angioplasty for the treatment of in-stent restenosis: a network meta-analysis of 11 randomized, controlled trials. JACC Cardiovasc Interv. 2015 Mar;8(3):382-394. doi: 10.1016/j.jcin.2014.09.023. Epub 2015 Feb 18. PMID 25703886
- [Result] Tank VH, Ghosh R, Gupta V, Sheth N, Gordon S, He W, Modica SF, Prestigiacomo CJ, Gandhi CD. Drug eluting stents versus bare metal stents for the treatment of extracranial vertebral artery disease: a meta-analysis. J Neurointerv Surg. 2016 Aug;8(8):770-4. doi: 10.1136/neurintsurg-2015-011697. Epub 2015 Jul 15. PMID 26180094
- [Result] Che WQ, Dong H, Jiang XJ, Peng M, Zou YB, Xiong HL, Yang YJ, Gao RL. Clinical outcomes and influencing factors of in-stent restenosis after stenting for symptomatic stenosis of the vertebral V1 segment. J Vasc Surg. 2018 Nov;68(5):1406-1413. doi: 10.1016/j.jvs.2018.02.042. Epub 2018 May 19. PMID 29789215
- [Result] Maciejewski DR, Pieniazek P, Tekieli L, Paluszek P, Przewlocki T, Tomaszewski T, Machnik R, Trystula M, Legutko J, Kablak-Ziembicka A. Comparison of drug-eluting and bare metal stents for extracranial vertebral artery stenting. Postepy Kardiol Interwencyjnej. 2019;15(3):328-337. doi: 10.5114/aic.2019.87887. Epub 2019 Sep 18. PMID 31592257
- [Result] Li J, Hua Y, Needleman L, Forsberg F, Eisenbray JR, Li Z, Liu R, Tian X, Jiao L, Liu JB. Arterial occlusions increase the risk of in-stent restenosis after vertebral artery ostium stenting. J Neurointerv Surg. 2019 Jun;11(6):574-578. doi: 10.1136/neurintsurg-2018-014243. Epub 2018 Oct 18. PMID 30337379
- [Result] Li L, Wang X, Yang B, Wang Y, Gao P, Chen Y, Zhu F, Ma Y, Chi H, Zhang X, Bai X, Feng Y, Dmytriw AA, Hong T, Hua Y, Jiao L, Ling F. Validation and comparison of drug eluting stent to bare metal stent for restenosis rates following vertebral artery ostium stenting: A single-center real-world study. Interv Neuroradiol. 2020 Oct;26(5):629-636. doi: 10.1177/1591019920949371. Epub 2020 Aug 16. PMID 32799746